CLINICAL TRIAL: NCT01088776
Title: Omega-3 Fatty Acid Supplementation to Treat Hypertriglyceridemia in Children With Chronic Kidney Disease
Brief Title: Omega-3 Fatty Acid Supplementation in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Elizabeth Harvey, Nephrologist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000012569
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease; Hypertriglyceridemia
Keywords: CKD; hypertriglyceridemia; Fatty Acid Supplementation; Children; Omega-3
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement (Experimental)
  Interventions: Dietary Supplement: n-3 Fatty Acid supplement
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n-3 Fatty Acid supplement — Children will be prescribed 1600-1800 mg EPA + DHA per m2 Body Surface Area, to a maximum of the upper limit of the age-appropriate range recommended by Health Canada.
  Each n-3FA gel capsule (1000 mg) will contain 400 mg EPA and 200 mg DHA derived from the oil of wild anchovies and sardines. A smaller gel capsule (500 mg; 200 mg EPA + 100 mg DHA) will be available for children unable to swallow large solid medication and a flavored liquid formulation, containing a similar proportion of EPA + DHA (2200 mg fish oil concentrate from anchovies and sardines, 750 mg EPA, 375 mg DHA per ½ teaspoon), will be available for use in toddlers and older children unable to swallow gel capsules.
  Arms: Supplement
Dietary Supplement: Placebo — The placebo, identical in opaque appearance and citrus-flavored taste, will contain a 50:50 blend of soybean and corn oil for both gel capsule (2 sizes) and liquid formulations.
  Arms: Control

SUMMARY:
Children with Chronic Kidney Disease (CKD) are at very high risk for cardiovascular morbidity and mortality. Hyper-lipidemia, a traditional risk factor for Cardiovascular Disease (CVD), occurs early in the progression of kidney failure; timely identification and intervention is prudent. Currently, there is no known effective therapy for hypertriglyceridemia, the most common lipid abnormality. n-3FA, in doses ranging from 2-6 g/day have effectively lowered elevated triglyceride (TG) levels by 20-50% in a variety of adult populations; however, their use in children with CKD has not been tested in a randomized controlled fashion. This study will provide important information on the safety, efficacy and tolerance of n-3FA in lowering elevated TG levels in children and adolescents with CKD.

DETAILED DESCRIPTION:
Following counseling on dietary and lifestyle changes to lower triglyceride levels, and a period of applying these modifications, children will be assigned in a random fashion to take either fish oil supplements or a placebo (soybean/corn oil) for 8 weeks. After this 8-week treatment period, children will not take a supplement for 4 weeks and then will be assigned the alternate product (fish oil or placebo) for another 8 weeks. Our main interest is to see whether there is a larger decrease in triglyceride levels after taking the fish oil supplement compared to the placebo.

The primary objective of this study is to determine whether omega-3 fatty acid supplements, given at therapeutic dosages over an 8-week period, significantly decrease elevated serum TG in children with CKD;

The secondary objectives of this study are:

i. To evaluate the effect of n-3 fatty acid supplements on total-, LDL-, and HDL-cholesterol;

ii. To determine whether n-3 fatty acid supplements are well tolerated by our study participants; and

iii. To test whether TG-lowering effects are sustained up to 4 weeks after stopping supplements.

ELIGIBILITY:
Inclusion Criteria:

* age at randomization: 2.0-17.4 years old (stratified by age: 2-8 yr, 9-13 yr, 14-17.4 yr)
* CKD stages 3 or 4 (GFR:15-59 ml/min/1.73 m2)
* established and stable in the CKD 3 and 4 Program for a minimum of 3 months
* fasting serum TG 95th percentile for age and gender 2 on more than or equal to 2 occasions

Exclusion Criteria:

* allergy to fish, corn, soybean
* anti-coagulant or anti-platelet drugs (heparin, warfarin, therapeutic NSAIDs) or herbal products (ginko, garlic, feverfew, ginger and ginseng) known to prolong bleeding
* currently undergoing treatment for dyslipidemia
* use of dietary supplements containing n-3FA
* children with Nephrotic Syndrome, on dialysis, or transplanted
* planned surgery, dialysis or transplantation within the next 7 months
* children with diabetes
* bleeding and clotting disorders:

  * thrombocytopenia (platelet count <100 x 109/L), including ITP, TTP
  * Von Willebrands disease
  * hemophilia
  * thrombophilia
  * vitamin K deficiency
  * severe liver disease
  * unstable patients with shock which can lead to DIC (disseminated intravascular coagulation)
  * active Henoch Schonlein Purpura
  * hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber disease)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Lipid Profiles(TG levels) | Week 1,4,12,16,24 and 28

SECONDARY OUTCOMES:
Platelet aggregation | Week 1,4,12,16,24 and 28
CBC | Week 1,4,12,16,24 and 28
Cholesterol Levels (LDL and HDL) | Week 1,4,12,16,24 and 28
Tolerability of n-3 fatty acid supplements by our participants | Week 1,4,12,16,24 and 28
  Sustainability of TG-lowering effects up to 4 weeks after stopping supplements

CONTACTS AND LOCATIONS:
Overall Officials: Donna Secker, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada